CLINICAL TRIAL: NCT01763099
Title: Mesenchymal Stem Cells Combined With Cord Blood for Treatment of Graft Failure Following Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Mesenchymal Stem Cells Combined With Cord Blood for Treatment of Graft Failure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Peking University People's Hospital (Other); Sun Yat-sen University (Other); Guangdong Provincial People's Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Southern Medical University, China (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFH-MSC-auto-HSCT-2013
Record Dates: First submitted 2013-01-05; First posted 2013-01-08 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Hematopoietic Stem Cell Transplantation; Mesenchymal Stem Cells; Umbilical Cord Blood; Graft Failure; Hematological Diseases
Keywords: Autologous Hematopoietic Stem Cell Transplantation; Mesenchymal Stem Cells; Cord Blood; Graft failure
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mesenchymal stem cells (Experimental): Mesenchymal stem cells group refers to treatment with mesenchymal stem cells (1×10^6 cells/kg, intravenously)
  Interventions: Biological: Mesenchymal stem cells
- Mesenchymal stem cells and cord blood (Experimental): Mesenchymal stem cells and cord blood group refers to treatment with mesenchymal stem cells (at a dose of 1×10^6 cells/kg) and cord blood
  Interventions: Biological: Mesenchymal stem cells and cord blood

INTERVENTIONS:
Biological: Mesenchymal stem cells — Mesenchymal stem cells will be intravenously infused via a central venous catheter(at a dose of 1×10^6 cells/kg, over 15 min) in day 1 and day 15 of the cycle. If the NEU and PLT levels do not attain the completely response(CR)standards after this cycle, mesenchymal stem cells combined with cord blood will be given. If the NEU and PLT levels attain the completely response(CR)or partly response(PR) standards after this cycle, another cycle with the same strategy will be given.
  Arms: Mesenchymal stem cells
Biological: Mesenchymal stem cells and cord blood — Mesenchymal stem cells will be given (at a dose of 1×10^6 cells/kg,intravenously infused via a central venous catheter)on day 1.day 15, day 29 and day 43 of the cycle. Cord blood will be given intravenously infused via a central venous catheter on day 2 of the cycle.
  Arms: Mesenchymal stem cells and cord blood

SUMMARY:
The purpose of this study is to evaluate the utility of treating patients experiencing graft failure after autologous hematopoietic stem cell transplantation with ex-vivo-expanded BM-drived mesenchymal stem cells from third-party donors or mesenchymal stem cells combined with cord blood. The first objective of this study was to evaluate the effect of such treatment on graft failure, and second object was to investigate the safety of such treatment.

DETAILED DESCRIPTION:
Autologous hematopoietic stem cell transplantation (auto-HSCT) are considered the standard of care for many malignancies, such as lymphoma, myeloma and some leukemias, and so on. Graft failure after auto-HSCT is a formidable complication. It occurs in 2-9.5% of patients and is associated with considerable morbidity and mortality related to infections and hemorrhagic complications. There are various options for the management of graft failure. The most common treatment of graft failure is growth factors such as granulocyte colony-stimulating factor (G-CSF)and recombinant erythropoietin,but it usually effective in the short term and no effect on platelet counts.

Mesenchymal stem cells (MSCs) are a form of multipotent adult stem cells that can be isolated from bone marrow (BM), adipose tissue, and cord blood. Clinical applications of human MSCs are evolving rapidly with goals of improving hematopoietic engraftment, preventing and treating graft-versus-host disease (GVHD) after allogeneic hematopoietic stem cell transplantation and so on.As an important source of hematopoietic stem cell, cord blood has been widely used in clinical practice. It is reported that cord blood combined with MSCs can increase engraftment after allogeneic hematopoietic stem cell transplantation. However, to our knowledge, the report about efficacy of treatment of graft that develops after auto-HSCT using expanded BM-derived MSCs from a third-party donor combined with cord blood is absent.If such treatment could be shown to be effective and safe, BM-derived MSCs could potentially be used as an universal donor material. This would have a major impact because the generation of donor-specific MSCs is time-consuming, costly, and often impractical if the clinical status of a patient is urgent.

In the present study, the investigators will prospectively evaluate the efficacy and safety of ex-vivo-expanded BM-derived MSCs from third-party donors or MSCs combined with cord blood in treating patients with graft failure after auto-HSCT.

ELIGIBILITY:
Inclusion Criteria:

* A patient age of 14-65 years
* Graft failure developing after auto-HSCT
* Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
* Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
hematopoietic recovery | 1 year
  Hematopoietic reconstitution post-transplantation is defined as reconstitution of both neutrophil and platelet numbers. Neutrophil reconstitution is defined as occurring on the first 3 consecutive days with an neutrophil(NEU)>0.5×10^9/L, and platelet (PLT) reconstitution is defined as the first >20×10^9/L for 3 consecutive days.

SECONDARY OUTCOMES:
infections, primary underlying disease relapse and any toxic side effects of MSCs treatment | 1 year
  Infections will be mainly focused within the first 100 days after MSCs treatment. Toxic side effects of treatment includes acute toxicity and late side effects. Acute toxicity principally involves the heart,live and kidney. Late toxic side effects involves principally the development of secondary tumors and relapse of the primary disease.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Koc ON, Lazarus HM. Mesenchymal stem cells: heading into the clinic. Bone Marrow Transplant. 2001 Feb;27(3):235-9. doi: 10.1038/sj.bmt.1702791. PMID 11277170
- [Background] Smith AR, Wagner JE. Alternative haematopoietic stem cell sources for transplantation: place of umbilical cord blood. Br J Haematol. 2009 Oct;147(2):246-61. doi: 10.1111/j.1365-2141.2009.07828.x. PMID 19796274